CLINICAL TRIAL: NCT05799664
Title: A Multicenter, Randomized, Single-blind, Sham-controlled Clinical Trial to Evaluate the Safety and Effectiveness of Targeted Lung Denervation Radiofrequency Ablation Devices in the Treatment of Chronic Obstructive Pulmonary Disease
Brief Title: Evaluation of Safety and Effectiveness of TLD Radiofrequency Ablation in the Treatment of COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Broncus Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-TLD-02
Record Dates: First submitted 2023-03-20; First posted 2023-04-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will be treated with TLD and standard of care (per GOLD guideline).
  Interventions: Device: TLD; Other: Standard of care
- Control group (Sham Comparator): Patients will undergo sham TLD procedure and be treated with standard of care (per GOLD guideline).
  Interventions: Other: Sham TLD procedure; Other: Standard of care

INTERVENTIONS:
Device: TLD — Patients allocated to experimental group will receive TLD therapy during which radiofrequency energy will be delivered to vagus nerve surrounding airway under bronchoscopy.
  Arms: Experimental group
Other: Sham TLD procedure — Patients allocated to control group will receive sham TLD procedure during which catheter will be placed in all treatment locations with no radiofrequency energy delivered.
  Arms: Control group
Other: Standard of care — Patients will also receive standard of care that meet the recommendations of GOLD guideline.

SUMMARY:
The objective of this trial is to evaluate the safety and effectiveness of Targeted Lung Denervation (TLD) for COPD patients using the lung denervation radiofrequency ablation device.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥40 and ≤ 75 years;
2. Diagnosis of COPD with post-bronchodilator PFT parameters FEV1/FVC<70% and 20% ≤ FEV1 ≤ 60% of predicted; if FEV1<30%pred, PaCO2≤50mmHg;
3. CAT ≥ 10 or mMRC ≥2;
4. Non-smoking for a minimum of 2 months prior to consent and agrees to not smoke for the duration of the clinical investigation;
5. Recent participation in a formal pulmonary rehabilitation program should have occurred ≥3 months prior to consent; if participants are currently enrolled in a maintenance program, they should agree to continue their current program through their 12-month follow-up visit;
6. Documented history of taking standard medication (consistent with GOLD guideline<2022>) for ≥12 months at the time of consent;
7. Received an influenza vaccine within the 12 months prior to consent or agrees to obtain an influenza vaccine during the clinical investigation, and agrees to annual influenza vaccines for the duration of the clinical investigation;
8. Resting SpO2 ≥ 89% at the time of screening;
9. Willing, able, and agrees to complete all protocol required baseline and follow-up testing assessments including finishing the Patient Diary;
10. Able to understand the purpose of the clinical investigation, agree to participate in the trial and able to complete the informed consent signature.

Exclusion Criteria:

1. BMI < 18 or > 35;
2. Asthma as defined by the GINA guideline (2022);
3. Patient has been previously diagnosed with a non-COPD active lung disease (e.g., active tuberculosis);
4. Patient has a medical history of pneumothorax;
5. Known contraindication or allergy to medications required for bronchoscopy or general anesthesia that cannot be medically controlled;
6. Recent respiratory infections or COPD exacerbation in preceding 4 weeks;
7. Malignancy treated with radiation or chemotherapy within 2 years of consent;
8. Daily use of > 10 mg of prednisone or its equivalent at the time of consent;
9. Recent (within 3 months of consent) opioid use;
10. Known gastrointestinal motility disorder or previous abdominal surgical procedure on stomach, esophagus, or pancreas
11. Has an implantable electronic device;
12. Previous or planned pulmonary or thoracic surgery (including but not limited to: pneumonectomy, lung transplantation, pulmonary medical device intervention < e.g. pulmonary valve implantation, bronchial thermal ablation (BT), etc. >) during this trial;
13. Myocardial infarction within last 6 months, EKG with evidence of life-threatening arrhythmias or acute ischemia, pre-existing documented evidence of a LVEF < 45%, stage C or D (ACC/AHA) or Class III or IV (NYHA) congestive heart failure, or any other cardiac findings that make the participant an unacceptable candidate for a bronchoscopic procedure utilizing general anesthesia;
14. High risk of pulmonary hypertension according to clinical assessment, defined as pulmonary artery systolic pressure estimated by echocardiogram to be > 50 mmHg;
15. Pulmonary nodule or other lesions thought to be at high risk of malignancy;
16. Clinically relevant bronchiectasis, defined as severe single lobe or multilobar bronchial wall thickening associated with airway dilation on CT scan leading to cough, intractable expectoration and repeated hemoptysis lasting for several days;
17. In the opinion of the Investigator, use of the TLD devices is not feasible, for example, due to screening chest CT scan reveals severe emphysema or bronchi anatomy cannot be fully treated with available catheter sizes: severe bullous disease (> 1/3 hemithorax) or site discovery of a mass that requires treatment;
18. A GCSI total symptom score ≥ 18.0 prior to treatment;
19. Any disease or condition that might interfere with completion of a procedure or this study (e.g., life expectancy< 1 years);
20. Women of childbearing potential must have a negative pregnancy test (blood or urine) pre-treatment and agree not to become pregnant for the duration of the study
21. Participated in any clinical trial and received experimental treatment within 3 months before the screening visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change of Forced expiratory volume in first second (FEV1) relative to baseline | 6 Months
  Defined as change in FEV1 at 6 months relative to baseline in the experimental group, compared to the control group.

SECONDARY OUTCOMES:
Time to first moderate or severe COPD exacerbation, first severe COPD exacerbation and first respiratory-related hospitalization. | 12 Months
  Defined as a comparison between study arms of the survival distributions for events based on log-rank tests.
Change in St. George's Respiratory Questionnaire COPD Version (SGRQ-C) Total score | 6 and 12 Months
  Defined as a comparison between study arms of the mean change in SGRQ-C from baseline.
  The SGRQ-C is a questionnaire developed to measure health status (quality of life) in COPD patients with a total and three component scores for: symptoms, activity and impacts; each score ranges from 0 (no impairment) to 100 (worst possible).
Change in modified Medical Research Council (mMRC) scale Total score | 6 and 12 Months
  Defined as a comparison between study arms of the mean change in mMRC from baseline.
  The modified Medical Research Council (mMRC) scale is recommended for conducting assessments of dyspnea and disability and functions. Total score ranging 0 to 4. The higher the score, the more deterioration in severity of dyspnea.
Change in COPD Assessment Test (CAT) Total score | 6 and 12 Months
  Defined as a comparison between study arms of the mean change in CAT from baseline.
  The CAT is a disease-specific HRQL with eight questions; each score ranges from 0 (no impairment) to 5 (worst possible). The CAT has a scoring range of 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Change in Pulmonary Function | 6 and 12 Months
  Defined as a comparison between study arms of the mean change in FEV1%pred, FVC(%pred), RV(%pred) from baseline.
Change in 6-minute walk distance (6MWD) | 6 and 12 Months
  Defined as a comparison between study arms of the mean change in 6MWD from baseline.
Device Success Rate of experimental group | Immediately after the procedure
  Defined as the proportion of the number of ablation procedures in which the catheter would be successfully placed on the treatment site and the catheter would be successfully withdrawn after the completion of the treatment procedure in all the ablation procedures.
(Serious) Adverse Event Rate related to device or procedure | Through study completion, an average of 1 year
  Defined as the total number of events per total number of treatment years.

CONTACTS AND LOCATIONS:
Overall Officials: Fengming Luo, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No